CLINICAL TRIAL: NCT01251289
Title: The Prevalence of Group B Streptococcus Positive Pregnant Patients in an Inner City Tertiary Care Center
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 09-072
Record Dates: First submitted 2010-11-30; First posted 2010-12-01 (Estimated); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Group B Streptococcus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
A retrospective review of the prevalence of Group B Streptococcus Positive Pregnant Patients in an Inner City Tertiary Care Center

DETAILED DESCRIPTION:
This is a retrospective chart review of the prevalence of Group B Streptococcus (GBS) positive patients

ELIGIBILITY:
Inclusion Criteria:

* GBS positive pregnant women

Exclusion Criteria:

* n/a

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Group B streptococcus positive pregnant women
Sampling Method: Probability Sample
Enrollment: 628 (Actual)
Dates: Start 2009-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Yudin, MD, Principal Investigator — Unity Health Toronto